CLINICAL TRIAL: NCT01196936
Title: Low-Dose Tamoxifen for Radiation-Induced Breast Cancer Risk Reduction: A Phase IIB Randomized Placebo-Controlled Trial
Brief Title: Low-Dose Tamoxifen Citrate in Reducing Breast Cancer Risk in Radiation-Induced Cancer Survivors
Acronym: LDTam
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH); St. Jude Children's Research Hospital (Other); University Health Network, Toronto (Other); University of Michigan (Other); Dana-Farber Cancer Institute (Other); Mayo Clinic (Other); University of Washington (Other); City of Hope National Medical Center (Other); M.D. Anderson Cancer Center (Other); University of Chicago (Other); University of Minnesota (Other); University of Colorado, Denver (Other); Wake Forest University (Other)
Responsible Party: Principal Investigator, Smitia Bhatia, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 08218; R01CA140245-01 (NIH); NCI-2010-01976 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-09-03; First posted 2010-09-09 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Cancer survivors; Low Dose Tamoxifen; Breast Cancer Risk Reduction
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Immunohistochemistry; Pharmacogenomic Testing; Biopsy, Fine-Needle

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (tamoxifen citrate) (Experimental): Patients receive tamoxifen citrate PO QD for 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Tamoxifen Citrate; Procedure: Digital mammography; Other: immunohistochemistry staining method; Other: pharmacological study; Other: laboratory biomarker analysis; Genetic: protein expression analysis; Other: pharmacogenomic studies; Other: questionnaire administration; Procedure: Fine needle aspiration; Other: Quality of Life Assessment
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO QD for 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Placebo; Procedure: Digital mammography; Other: immunohistochemistry staining method; Other: pharmacological study; Other: laboratory biomarker analysis; Genetic: protein expression analysis; Other: pharmacogenomic studies; Other: questionnaire administration; Procedure: Fine needle aspiration; Other: Quality of Life Assessment

INTERVENTIONS:
Drug: Tamoxifen Citrate — 5 mg PO Daily
  Other Names: Marketed under trade name Nolvadex as 10 mg and 20 mg tablets; ICI 46,474
  Arms: Arm I (tamoxifen citrate)
Drug: Placebo — 1 tablet daily
  Arms: Arm II (placebo)
Procedure: Digital mammography — Correlative studies
Other: immunohistochemistry staining method — Correlative Studies
Other: pharmacological study — Correlative Studies
Other: laboratory biomarker analysis — Correlative Studies
Genetic: protein expression analysis — correlative studies
Other: pharmacogenomic studies — correlative studies
Other: questionnaire administration — Ancillary studies
Procedure: Fine needle aspiration
  Other Names: Correlative studies
Other: Quality of Life Assessment — Ancillary Studies

SUMMARY:
Estrogen can cause the growth of breast cancer cells. Hormone therapy using tamoxifen citrate may fight breast cancer by blocking the use of estrogen by the tumor cells

This phase IIb trial studies how well low-dose tamoxifen citrate works in reducing breast cancer risk in radiation-induced cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the impact of a two-year course of low-dose tamoxifen (tamoxifen citrate) administered at 5 mg per day on surrogate endpoint biomarkers of breast cancer (BC) risk, including: mammographic breast density (MBD), an established radiographic biomarker of BC risk; cytomorphology and proliferative index, tissue biomarkers closely linked to BC risk; and sex steroid hormones and insulin growth factors, circulating biomarkers of BC risk.

II. To establish safety and tolerability of this low-dose tamoxifen regimen, assessing both objective measures (lipid profiles, clotting factors and bone metabolism markers) and patient-reported outcomes.

III. To examine the modifying effect of demographic, clinical, and molecular characteristics on the risk: benefit ratio from this two-year low dose tamoxifen intervention.

IV. To explore the relationship between this low-dose tamoxifen regimen and clinical measures of efficacy (new breast cancer and ductal carcinoma in situ [DCIS] diagnoses) and toxicity (thromboembolic events, reports of hot flashes and gynecological symptoms, liver function abnormalities, and other cancer diagnoses).

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive tamoxifen citrate orally (PO) once daily for 24 months in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive placebo PO once daily for 24 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Exposure to radiation therapy (RT) delivered to the chest, axilla, and/or supraclavicular areas at a cumulative dose of 12 Gy or more by age 40 years; in addition, patients who received total body irradiation by age 40 may be considered
* No evidence of active disease from their primary cancer for at least 2 continuous years prior to registration; the indication for RT is not specified but cannot be for primary breast cancer; common examples include, but are not limited to: lymphoma, leukemia, sarcoma, and Wilms tumor occurring in pediatric patients, and lymphoma, leukemia, and sarcoma occurring in young adults; primary cancer therapy must have been completed at least 6 months prior to registration
* Well-defined menopausal status falling into one of the following categories:

  * Premenopausal, defined as age at registration 45 years old or younger with regular monthly period for at least 6 consecutive months prior to registration
  * Postmenopausal, defined as continuous absence of menstruation for 12 months OR status-post bilateral oophorectomy OR follicle stimulating hormone (FSH) level in the postmenopausal range

Exclusion Criteria:

* Subsequent malignant neoplasm (SMN) other than those listed below diagnosed within 2 years of study entry; patients with the listed indolent or pre-invasive neoplasms may be eligible if diagnosed within 2 years and all treatment was completed at least 6 months prior to registration:

  * Non-melanoma cancers of the skin
  * Thyroid cancer
  * Cervical cancer confined to the cervix or cervical intraepithelial neoplasia (CIN)
  * Ductal carcinoma in situ (DCIS) or breast intraepithelial neoplasia (IEN) (includes atypical hyperplasia and lobular carcinoma in situ [LCIS]), or
  * Superficial or non-invasive transitional cell carcinoma of the bladder
* For women with a prior history of DCIS or breast IEN, only one breast could have been involved and all therapy must have been completed at least 6 months prior to registration; in addition women with a prior history of invasive breast cancer may also be eligible, as long as only one breast was involved, they were diagnosed at least 2 years prior to study entry, and therapy was completed at least 6 months prior to study entry
* Bilateral breast implants or status-post bilateral prophylactic mastectomy
* Evidence of malignant breast disease on any form of breast imaging; the study only requires annual mammography; however, annual breast magnetic resonance imaging (MRI) is considered standard of care in this patient population (per Children's Oncology Group [COG] or National Comprehensive Cancer Network [NCCN] follow-up guidelines), and breast ultrasound may be indicated if a palpable lesion is detected on screening clinical breast exam; abnormal imaging may require additional radiographs and/or breast biopsy; patients who are found to have benign breast disease with or without atypia may continue on study as long as there is no evidence of malignancy; if there is evidence of malignancy, and only one breast is involved, they may be reapproached 6 months after completion of therapy for consideration of the trial
* Baseline categorical mammographic density scored as BIRAD 1, or extremely fatty, in both breasts; if the patient has a prior history of IEN (DCIS, LCIS, or atypical hyperplasia), the contralateral breast must not have a mammographic density score of BIRAD 1; this determination will be made at the local site
* Current or recent use (within 6 months of registration or baseline mammogram, whichever is first) of any of the following: systemic hormone replacement therapy (includes oral or transdermal formulations); Vagifem and Estring, two formulations of locally applied vaginal estrogen associated with minimal systemic absorption, may be allowed; other estrogen-containing vaginal creams, while not an exclusion, should be avoided whenever possible; patients with a history of hormone modifying herbal supplements are eligible, but patients will be asked to avoid their use after on study
* Current or recent use (within 6 months of registration or baseline mammogram, whichever is first) of any of the following: hormonal forms of contraception (includes oral, transdermal, implanted, and injectable formulations): selective estrogen receptor modifiers; aromatase inhibitors; GnRH analogs; androgens or antiandrogens
* Concurrent use of warfarin and strong inhibitors or CYP2D6 will not be allowed
* A personal history or a strong family of thromboembolism, including deep venous thrombosis (DVT), pulmonary embolus (PE), or cerebrovascular accident (CVA); a personal history of transient ischemic attack (TIA) or retinal vein thrombosis will also not be allowed; in addition, patients with a condition known to increase hypercoagulability, such as Factor V Leiden disease, will be excluded; patients with atrial fibrillation will be excluded, due to risk of CVA, but patients with coronary artery disease or congestive heart failure without atrial fibrillation will be allowed to participate
* Current intrauterine pregnancy or plans to become pregnant within two years; in addition, currently nursing mothers will be excluded
* Serum creatinine > 2X the institutional norm
* Total bilirubin > 2X the institutional norm
* Serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic pyruvic transaminase (SGPT) > 2X the institutional norm
* Unable to provide consent

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-09; Primary Completion 2018-12-11 (Actual); Study Completion 2028-12-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Smita Bhatia, MD, Principal Investigator — University of Alabama at Birmingham
Locations (13):
- United States (12):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope Medical Center, Duarte, California
  - University of Colorado, Anschutz Medical Campus, Aurora, Colorado
  - University of Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Wake Forest University, Winston-Salem, North Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - MD Anderson, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
- University Health Network, Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened for eligibility at each participating institution.However, after central review of mammograms, 11 participants were ineligible for the study (mammographic density <25%) and 1 participant was randomized but withdrew before taking the study drug. These 12 participants were excluded from the analysis.
Groups:
- Arm I (Tamoxifen Citrate): Patients receive tamoxifen citrate PO QD for 24 months in the absence of disease progression or unacceptable toxicity.
  Tamoxifen Citrate: 5 mg PO Daily
  Digital mammography: Correlative studies
  immunohistochemistry staining method: Correlative Studies
  pharmacological study: Correlative Studies
  laboratory biomarker analysis: Correlative Studies
  protein expression analysis: correlative studies
  pharmacogenomic studies: correlative studies
  questionnaire administration: Ancillary studies
  Fine needle aspiration
  Quality of Life Assessment: Ancillary Studies
- Arm II (Placebo): Patients receive placebo PO QD for 24 months in the absence of disease progression or unacceptable toxicity.
  Placebo: 1 tablet daily
  Digital mammography: Correlative studies
  immunohistochemistry staining method: Correlative Studies
  pharmacological study: Correlative Studies
  laboratory biomarker analysis: Correlative Studies
  protein expression analysis: correlative studies
  pharmacogenomic studies: correlative studies
  questionnaire administration: Ancillary studies
  Fine needle aspiration
  Quality of Life Assessment: Ancillary Studies
Period: Overall Study
Arm/Group | Arm I (Tamoxifen Citrate) | Arm II (Placebo)
Started | 34 | 38
Year one post treatment | 27 | 28
Completed | 23 | 21
Not Completed | 11 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Tamoxifen Citrate) | Arm II (Placebo) | Total
Number analyzed (Participants) | 34 | 38 | 72
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 43.7 [34.3 to 48.8] | 44.1 [34.6 to 47.0] | 43.8 [34.5 to 48.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 38 | 72
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 31 | 33 | 64
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 30 | 36 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 2 | 3
  United States | 33 | 36 | 69

OUTCOME MEASURES:

1. Primary Outcome: Mammographic Breast Density
Description: Mammographic density was quantified as percentage of fibroglandular tissue. Using an intention-to-treat analysis, mammographic breast density (MBD) was compared between patients in the low dose tamoxifen intervention and placebo group by applying the linear mixed effects model for normally distributed data.
Time Frame: At year two post treatment
Measure: Least Squares Mean (Standard Error); unit: percentage of fibrogladular tissue
Arm/Group | Arm I (tamoxifen citrate) | Arm II (placebo)
Number analyzed (Participants) | 23 | 21
percentage of fibrogladular tissue | 45.2 (2.4) | 48.6 (2.5)
Statistical Analysis 1: Comparison: Arm I (tamoxifen citrate) vs Arm II (placebo); Test type: Superiority; p = 0.05, Mixed Models Analysis — The calculated p-value is 0.05

2. Secondary Outcome: Insulin Growth Factor Levels (IGF1)
Description: IGF1 will be treated as a continuous measure. The linear mixed effects model for between group comparisons of measures from 3 time points will be applied. The unstructured mean model and linear in time model will be employed.
Time Frame: Up to 2 years
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Arm I (tamoxifen citrate) | Arm II (placebo)
Number analyzed (Participants) | 34 | 38
ng/mL | 144.3 (7.1) | 162.3 (7.2)
Statistical Analysis 1: Comparison: Arm I (tamoxifen citrate) vs Arm II (placebo); Test type: Superiority; p = 0.0266, Mixed Models Analysis

3. Secondary Outcome: Number of Grade 2-4 Toxicities
Description: Will be tabulated by treatment arm. Differences by treatment arm will be evaluated using Fisher exact tests.
Time Frame: Up to 2 years
Measure: Number; unit: Adverse Events
Arm/Group | Arm I (tamoxifen citrate) | Arm II (placebo)
Number analyzed (Participants) | 34 | 38
Adverse Events | 77 | 40
Statistical Analysis 1: Comparison: Arm I (tamoxifen citrate) vs Arm II (placebo); Test type: Superiority; p = 0.12, Fisher Exact

4. Secondary Outcome: Biomarker Levels
Description: Total cholesterol, low and high density lipoprotein, triglycerides, and anti-thrombin III enzymatic assay measurements will be treated as continuous variables. Transformed to normality as appropriate, the linear mixed effects model will be applied, using the unstructured mean model and linear in time model to assess the effects of low-dose tamoxifen on these measurements over time.
Time Frame: Up to 2 years
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Arm I (tamoxifen citrate) | Arm II (placebo)
Number analyzed (Participants) | 34 | 38
mg/dL
  Total Cholesterol | 189.9 (7.1) | 192.5 (7.2)
  Low-density lipoprotein | 105.4 (5.7) | 108.6 (5.8)
  High-density lipoprotein | 57.6 (3.0) | 56.5 (3.0)
  Triglycerides | 138.1 (13.2) | 116.6 (13.5)
  Anti-thrombin III | 89.3 (5.4) | 98.1 (5.7)
Statistical Analysis 1: Comparison: Arm I (tamoxifen citrate) vs Arm II (placebo); Test type: Superiority; p > 0.05, Mixed Models Analysis

5. Secondary Outcome: Percentage of Pills Taken Out of the Total Prescribed
Description: The number of pills taken out of the total prescribed in a 3-month period will be modeled as a random effects binomial regression model. The binomial rates from 8 time points (month 3-24) will be modeled as unstructured mean model with 7 indicator variables as well as polynomial models over time. The random-intercept and the random intercept and slope models will be considered. The significance of the time indicators or parameters by treatment interaction will be evaluated for treatment difference in compliance.
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: percentage of pills taken
Arm/Group | Arm I (tamoxifen citrate) | Arm II (placebo)
Number analyzed (Participants) | 34 | 38
percentage of pills taken | 97.5 [56.1 to 100] | 96.7 [20.7 to 99.9]
Statistical Analysis 1: Comparison: Arm I (tamoxifen citrate) vs Arm II (placebo); Test type: Superiority; p = 0.78, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Number of Participants With Different Patient Reported Symptoms, Measured by Questionnaire
Description: The outcomes will be scored as a 5-point Likert-type scale (0-4) in response to questions on how much the patients are bothered by certain symptoms. The questionnaire will be administered every 6 months. The responses will be treated as normally distributed, as ordinal or dichotomized variable, and the linear mixed effects of general linear mixed model (GLMM) methods will be applied to compare changes between treatment groups. Piecewise models will also be fitted with join point at 6 months, considering linear and curvilinear trajectories between 6 and 24 month time points.
Time Frame: Up to 2 years
Population: Symptoms with >10% prevalence are reported; patients were dichotomized into 2 groups: those that rated the symptom as moderately or extremely bothersome vs. slightly or quite a bit bothersome
Measure: Number; unit: participants
Arm/Group | Arm I (tamoxifen citrate) | Arm II (placebo)
Number analyzed (Participants) | 34 | 38
participants
  Interrupted sleep | 16 | 16
  General aches or pains | 14 | 8
  Hot flashes | 13 | 12
  Joint pain or stiffness | 12 | 9
  Feeling unusually tired | 12 | 10
  Heartburn and/or acid stomach | 11 | 10
  Headaches | 11 | 14
  Muscle cramps or soreness | 11 | 8
Statistical Analysis 1: Comparison: Arm I (tamoxifen citrate) vs Arm II (placebo); Test type: Superiority; p > 0.05, Chi-squared

7. Secondary Outcome: Insulin Growth Factor Levels (IGF3 )
Description: IGF3 will be treated as a continuous measure. The linear mixed effects model for between group comparisons of measures from 3 time points will be applied. The unstructured mean model and linear in time model will be employed.
Time Frame: Up to 2 years
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Arm I (tamoxifen citrate) | Arm II (placebo)
Number analyzed (Participants) | 34 | 38
ng/mL | 4716.0 (168.0) | 4315.2 (170.8)
Statistical Analysis 1: Comparison: Arm I (tamoxifen citrate) vs Arm II (placebo); Test type: Superiority; p = 0.071, Mixed Models Analysis

8. Secondary Outcome: Biomarker Levels - Alkaline Phosphatase
Description: Serum bone-specific alkaline phosphatase measurements will be treated as continuous variables. Transformed to normality as appropriate, the linear mixed effects model will be applied, using the unstructured mean model and linear in time model to assess the effects of low-dose tamoxifen on these measurements over time.
Time Frame: Up to 2 years
Measure: Least Squares Mean (Standard Error); unit: ug/L
Arm/Group | Arm I (tamoxifen citrate) | Arm II (placebo)
Number analyzed (Participants) | 34 | 38
ug/L | 12.2 (0.7) | 12.4 (0.7)
Statistical Analysis 1: Comparison: Arm I (tamoxifen citrate) vs Arm II (placebo); Test type: Superiority; p = 0.739, Mixed Models Analysis

9. Secondary Outcome: Biomarker Levels - Urine N-telopeptide
Description: Urine n-telopeptide measurements will be treated as continuous variables. Transformed to normality as appropriate, the linear mixed effects model will be applied, using the unstructured mean model and linear in time model to assess the effects of low-dose tamoxifen on these measurements over time.
Time Frame: Up to 2 years
Measure: Least Squares Mean (Standard Error); unit: nM Bone Collagen Equiv. / nM Creatinine
Arm/Group | Arm I (tamoxifen citrate) | Arm II (placebo)
Number analyzed (Participants) | 34 | 38
nM Bone Collagen Equiv. / nM Creatinine | 33.1 (3.6) | 32.0 (3.8)
Statistical Analysis 1: Comparison: Arm I (tamoxifen citrate) vs Arm II (placebo); Test type: Superiority; p = 0.8315, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse events were collected every six months while the participants were on the two year study.
Arm/Group | Arm I (Tamoxifen Citrate) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/38
Serious Adverse Events (participants affected / at risk) | 2/34 | 3/38
Other Adverse Events (participants affected / at risk) | 26/34 | 25/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Tamoxifen Citrate) (N=34) | Arm II (Placebo) (N=38)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Tamoxifen Citrate) (N=34) | Arm II (Placebo) (N=38)
Hot flashes (Vascular disorders) | 8 | 10
Weight loss (Investigations) | 7 | 8
Weight gain (Investigations) | 9 | 7
Psychiatric disorders - Other (Psychiatric disorders) | 9 | 7 — Mood swings, Unhappy with body appearance
Depression (Psychiatric disorders) | 7 | 7
Insomnia (Psychiatric disorders) | 4 | 7
Irregular menstruation (Reproductive system and breast disorders) | 8 | 6
Headache (Nervous system disorders) | 8 | 6
Endrocrine disorders - Other (Endocrine disorders) | 6 | 6 — Night sweats
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 6
Dry mouth (Gastrointestinal disorders) | 3 | 6
Diarrhea (Gastrointestinal disorders) | 6 | 5
Breast pain (Reproductive system and breast disorders) | 6 | 5
Constipation (Gastrointestinal disorders) | 6 | 5
Malaise (General disorders) | 6 | 5
Dizziness (Nervous system disorders) | 5 | 5
Reproductive system and breast disorders-Other (Reproductive system and breast disorders) | 5 | 6 — Vaginal dryness, vaginal spotting, genital itching/irritation
Gastrointestinal disorders - other (Gastrointestinal disorders) | 5 | 5 — Increased appetite, decreased appetite
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 5
Irritability (General disorders) | 5 | 5
Vaginal Hemorrhage (Reproductive system and breast disorders) | 4 | 5
Blurred vision (Eye disorders) | 3 | 5
Nausea (Gastrointestinal disorders) | 3 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 5
Urinary frequency (Renal and urinary disorders) | 1 | 5
Somnolence (Nervous system disorders) | 8 | 4
Vaginal discharge (Reproductive system and breast disorders) | 8 | 4
Restlessness (Psychiatric disorders) | 6 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Gastroesophageal reflux disease (Gastrointestinal disorders) | 6 | 4
Urinary incontinence (Renal and urinary disorders) | 5 | 4
Bloating (Gastrointestinal disorders) | 4 | 4
Palpitations (Cardiac disorders) | 3 | 4
General disorders - Other (General disorders) | 11 | 3 — Fluid retention, intolerance of cold, intolerance of heat
Fatigue (General disorders) | 10 | 3
Nervous system disorders - Other (Nervous system disorders) | 9 | 3 — Easily distracted, clumsiness
Bruising (Injury, poisoning and procedural complications) | 8 | 3
Concentration impairment (Nervous system disorders) | 7 | 3
Non-cardiac chest pain (General disorders) | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Paraesthesia (Nervous system disorders) | 6 | 2
Memory impairment (Nervous system disorders) | 6 | 2
Flatulence (Gastrointestinal disorders) | 3 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 2
Cystitis noninfective (Renal and urinary disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 1
Tremor (Nervous system disorders) | 4 | 1
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Agitation (Psychiatric disorders) | 2 | 1
Dyspareunia (Reproductive system and breast disorders) | 4 | 0
Renal and urinary disorders - Other (Renal and urinary disorders) | 2 | 0 — burning upon urination; strong urine smell
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2 | 0 — Leg cramps
Pelvic pain (Reproductive system and breast disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Slower than expected accrual, and financial constraints of supporting the study drug costs necessitated study closure before attainment of planned study enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-26): https://cdn.clinicaltrials.gov/large-docs/36/NCT01196936/Prot_SAP_000.pdf